CLINICAL TRIAL: NCT06442592
Title: CATAMARAN - Pediatrics : Characterization and Support for Neurodevelopmental Disorders Associated with Congenital Heart Defects
Brief Title: Characterization and Support for Neurodevelopmental Disorders Associated with Congenital Heart Defects
Acronym: CATAMARAN Ped
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: University of Angers - Pays de la Loire psychology laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RC23_0548; 2024-A00428-39 (Other: ANSM (IDRCB))
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Congenital Heart Defects; Neurodevelopmental Disorder
Keywords: Congenital Heart Defects; Neurodevelopmental Disorder; Genetics
MeSH Terms: conditions — Heart Defects, Congenital; Neurodevelopmental Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CATAMARAN - Pediatrics - Nantes (Other): The study population will consist of 201 children aged 3 to 11 and their two parents.
  Interventions: Other: Blood sampling; Diagnostic Test: Assessment of neurodevelopment (Nantes); Other: Assessment of the parental stress
- CATAMARAN - Pediatrics - Associated centers (excluding Nantes) (Other): The study population will consist of 201 children aged 3 to 11 and their two parents.
  Interventions: Other: Blood sampling; Diagnostic Test: Assessment of neurodevelopment (CA); Other: Assessment of the parental stress

INTERVENTIONS:
Other: Blood sampling — An EDTA blood sample will be taken from the children and their two parents. Sample volume will be 2 x 3mL.
Diagnostic Test: Assessment of neurodevelopment (CA) — The children will be seen by a neuropsychologist, who will then determine whether or not they have neurodevelopmental disorders.
  Arms: CATAMARAN - Pediatrics - Associated centers (excluding Nantes)
Diagnostic Test: Assessment of neurodevelopment (Nantes) — The children will be seen by a multidisciplinary team (including a neuropsychologist), who will then determine whether or not they have neurodevelopmental disorders.
  Arms: CATAMARAN - Pediatrics - Nantes
Other: Assessment of the parental stress — Parents' parental stress will be assessed using the Parental Stress Index (PSI) questionnaire.

SUMMARY:
The leading cause of birth defects, Congenital Heart Defects (CHD) affect 12 million people worldwide and 41,000 newborns/year in Europe. It's a major cause of life-long morbidity and mortality, and a crucial public health issue. More than 50% of childs born with critical CHD will develop Neurodevelopmental Disorders (NDs), requiring specific care and impairing quality of life. NDs corresponds to early and lasting disturbances in cognitive, affective and behavioral development, linked to abnormalities in brain development. They are heterogeneous, affecting language, learning, motor skills, intellectual efficiency, social cognition, attention, memory and executive functions, and are associated with psychosocial difficulties (adaptive behavior, social interactions). This hidden handicap is the main long-term sequels of CHD, even before cardiovascular sequels, in individuals who often underwent multiple heart operations in early childhood. NDs concern not only complex CHD, but also simple CHD repaired in childhood and considered cured.

The origin of TND associated with CHD is largely unknown. To date, few genetic or environmental causes have been clearly identified, but recent work has suggested that a common origin may link cardiac malformation and neurodevelopmental abnormality.

The CATAMARAN - Pediatrics project is designed to detect potential neurodevelopmental delays associated with CHD as early as age 3, and to identify individual susceptibility factors involved in the occurrence of NDs in CHD children.

ELIGIBILITY:
Inclusion Criteria:

* Child (aged 3 to 11) with critical MCC operated on for heart surgery during the first three months of life
* Parents and child affiliated with or benefiting from a social security or similar scheme
* Parents' and child's good understanding of the French language
* Free, informed and written consent of both parents for themselves and for the child
* Free, informed and written consent of the child aged 6 and over
* Biological parents

Exclusion Criteria:

* Genetic anomaly or malformative syndrome associated with neurodevelopmental abnormalities, identified prior to inclusion
* Neurodevelopmental assessment not practicable

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1206 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of the prevalence of neurodevelopmental disorders in children aged 3-11 years with critical congenital heart defects. | 14 days

SECONDARY OUTCOMES:
Identify rare genetic variants associated with genome-wide neurodevelopmental disorders in patients with congenital heart defects. | One day
  The presence of rare genetic variants associated with neurodevelopmental disorders will be determined by a 30X whole genome sequencing approach based on the association study of congenital heart defects with neurodevelopmental disorders versus congenital heart defects without neurodevelopmental disorders.
Identify frequent genetic variants associated with genome-wide neurodevelopmental disorders in patients with congenital heart defects. | One day
  The presence of frequent genetic variants associated with neurodevelopmental disorders will be determined by a 30X whole genome sequencing approach based on the association study of congenital heart defects with neurodevelopmental disorders versus congenital heart defects without neurodevelopmental disorders.
Assessment of the prevalence of neurodevelopmental disorders in children with critical congenital heart defects in each age subgroup (3-5, 6-8, and 9-11 years). | up to 14 days
Evaluate and describe the neurodevelopmental domains affected in the pediatric population of Nantes. | up to 14 days
  Functional diagnosis of different types of NDD defined by at least one score deficient in relation to the test norm (-1.5 standard deviation or 90 percentile) in each age subgroup.
Assessment of the quality of life and psychopathological aspects of the child as well as parental stress. | up to 14 days
  Proportion of children with impaired quality of life, psychopathological difficulties and proportion of adults with parental stress, compared with the test norm (-1.5 standard deviation or 90 percentile).
Assessment of diagnostic accuracy (of NDD) provided by an innovative multidisciplinary approach. | up to 14 days
  Comparison of TND frequency in Nantes versus associated centers and description of differences between centers
Describe the different types of neurodevelopmental disorders (number and nature of neurodevelopmental domains affected) in each age subgroup (intelligence, oral language, motor skills, school learning, executive functions, social interactions). | up to 14 days

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Chu Brest, Brest, Brittany Region
  - CHU Rennes, Rennes, Brittany Region
  - CHU Nantes, Nantes, Loire-Atlantique
  - CHU Angers, Angers, Maine-et-Loire
  - CHU Tours, Tours, Val de Loire

IPD SHARING:
Plan to Share IPD: Undecided